CLINICAL TRIAL: NCT00619177
Title: Assessing the Impact of MOVALIS on Health Related Quality of Life
Brief Title: Assessing the Impact of MOVALIS in Osteoarthritis and Rheumatoid Arthritis Patients on Health Related Quality of Life
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 107.273
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Results first posted 2009-11-18 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: Osteoarthritis; Arthritis, Rheumatoid
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The objective of the observational study is to examine the effect of MOVALIS (Meloxicam) therapy on Health Related Quality of Life (HRQoL) in the diverse region of Central and Eastern Europe. The Medical Outcomes Study 12 Item Short Form Health Survey version 2 (SF-12v2) will be used as the instrument to measure any change in physical wellbeing (Physical Component Summary, PCS) and mental wellbeing (Mental Component Summary, MCS) of patients following MOVALIS (Meloxicam) therapy.

ELIGIBILITY:
Inclusion Criteria (according to Summary of Product Characteristics (SPC) ):

1. Male or female patients aged 18 years or above 2 Females of child bearing age must be using adequate contraception (hormonal or barrier method of birth control) 3. Patients with symptoms of acute, painful osteoarthritis or rheumatoid arthritis 4. Patients requiring therapy with non-steroidal anti-inflammatory drugs (NSAIDs) 5. Patients requiring either parenteral and/or oral NSAIDs 6. Patients who have not taken another NSAID or Cyclo-oxygenase-2 (COX-2) inhibitor in the previous 7 days Pain intensity on the visual analogue scale (VAS) 25 mm and above

Exclusion Criteria (according to contraindications of Summary of Product Characteristics (SPC) ):

1. Known hypersensitivity to meloxicam or any excipient of the product, known or suspected hypersensitivity to analgesics, antipyretics or NSAIDs
2. Patients who have developed signs of asthma, nasal polyps, angio-oedema or urticaria following the administration of aspirin or other NSAIDs
3. Active peptic ulcer, gastrointestinal perforation or bleeding within the last 6 months
4. Severe liver failure
5. Non-dialysed severe renal failure
6. Pregnancy or breastfeeding
7. Haemostasis disorders or concomitant treatment with anticoagulants
8. Severe congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care and rheumatology clinics
Sampling Method: Non-Probability Sample
Enrollment: 3569 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (319):
- Croatia (2):
  - Boehringer Ingelheim Investigational Site, Split
  - Boehringer Ingelheim Investigational Site, Zagreb
- Czechia (253):
  - Boehringer Ingelheim Investigational Site, Aš
  - Boehringer Ingelheim Investigational Site, Babice
  - Boehringer Ingelheim Investigational Site, Benátky nad Jizerou
  - Boehringer Ingelheim Investigational Site, Benesov Nad Ploucnicí
  - Boehringer Ingelheim Investigational Site, Benesov U Prahy
  - Boehringer Ingelheim Investigational Site, Benešov
  - Boehringer Ingelheim Investigational Site, Beroun
  - Boehringer Ingelheim Investigational Site, Bílina
  - Boehringer Ingelheim Investigational Site, Bílovec
  - Boehringer Ingelheim Investigational Site, Bílovice nad Svitavou
  - Boehringer Ingelheim Investigational Site, Blansko
  - Boehringer Ingelheim Investigational Site, Blatnice pod Svatým Antonínkem
  - Boehringer Ingelheim Investigational Site, Bohusovice Nad Ohrí
  - Boehringer Ingelheim Investigational Site, Bolatice
  - Boehringer Ingelheim Investigational Site, Boskovice
  - Boehringer Ingelheim Investigational Site, Bratríkov
  - Boehringer Ingelheim Investigational Site, Brno
  - Boehringer Ingelheim Investigational Site, Broumov
  - Boehringer Ingelheim Investigational Site, Bruntál
  - Boehringer Ingelheim Investigational Site, Břeclav
  - Boehringer Ingelheim Investigational Site, Buchlovice
  - Boehringer Ingelheim Investigational Site, Bystřice nad Pernštejnem
  - Boehringer Ingelheim Investigational Site, Byšice
  - Boehringer Ingelheim Investigational Site, Cáslav
  - Boehringer Ingelheim Investigational Site, Ceská Lípa
  - Boehringer Ingelheim Investigational Site, Ceská Trebová
  - Boehringer Ingelheim Investigational Site, Ceské Budojovice
  - Boehringer Ingelheim Investigational Site, Ceský Tesín
  - Boehringer Ingelheim Investigational Site, Cheb
  - Boehringer Ingelheim Investigational Site, Chodov
  - Boehringer Ingelheim Investigational Site, Chomutov
  - Boehringer Ingelheim Investigational Site, Chropyně
  - Boehringer Ingelheim Investigational Site, Chrudim
  - Boehringer Ingelheim Investigational Site, Černošice
  - Boehringer Ingelheim Investigational Site, Černožice
  - Boehringer Ingelheim Investigational Site, Decín
  - Boehringer Ingelheim Investigational Site, Dobrís
  - Boehringer Ingelheim Investigational Site, Dobruška
  - Boehringer Ingelheim Investigational Site, Dobřany
  - Boehringer Ingelheim Investigational Site, Dol . Lou.
  - Boehringer Ingelheim Investigational Site, Dolní Benesov
  - Boehringer Ingelheim Investigational Site, Dolní Berkovice
  - Boehringer Ingelheim Investigational Site, Domažlice
  - Boehringer Ingelheim Investigational Site, Drnovice
  - Boehringer Ingelheim Investigational Site, Dvur Králové Nad Labem
  - Boehringer Ingelheim Investigational Site, Frenstát
  - Boehringer Ingelheim Investigational Site, Fryštát
  - Boehringer Ingelheim Investigational Site, Frýdek-Místek
  - Boehringer Ingelheim Investigational Site, Frýdlant
  - Boehringer Ingelheim Investigational Site, Fulnek
  - Boehringer Ingelheim Investigational Site, Hanušovice
  - Boehringer Ingelheim Investigational Site, Havírov
  - Boehringer Ingelheim Investigational Site, Havlíckuv Brod
  - Boehringer Ingelheim Investigational Site, Heřmanův Městec
  - Boehringer Ingelheim Investigational Site, Hlucín
  - Boehringer Ingelheim Investigational Site, Hluk
  - Boehringer Ingelheim Investigational Site, Hodonice
  - Boehringer Ingelheim Investigational Site, Hodonín
  - Boehringer Ingelheim Investigational Site, Holešov
  - Boehringer Ingelheim Investigational Site, Holice
  - Boehringer Ingelheim Investigational Site, Horice V Podkrkonosí
  - Boehringer Ingelheim Investigational Site, Horní Berkovice
  - Boehringer Ingelheim Investigational Site, Horní Slavkov
  - Boehringer Ingelheim Investigational Site, Hořovice
  - Boehringer Ingelheim Investigational Site, Hostinné
  - Boehringer Ingelheim Investigational Site, Hošťka
  - Boehringer Ingelheim Investigational Site, Hradec Králové
  - Boehringer Ingelheim Investigational Site, Hrádek n.N.
  - Boehringer Ingelheim Investigational Site, Hronov
  - Boehringer Ingelheim Investigational Site, Hrušovany nad Jevišovkou
  - Boehringer Ingelheim Investigational Site, Hulín
  - Boehringer Ingelheim Investigational Site, Hustopece U Brna
  - Boehringer Ingelheim Investigational Site, Hustopeče
  - Boehringer Ingelheim Investigational Site, Jablonec
  - Boehringer Ingelheim Investigational Site, Jablonec n.N.
  - Boehringer Ingelheim Investigational Site, Jablunkov
  - Boehringer Ingelheim Investigational Site, Jaroměř
  - Boehringer Ingelheim Investigational Site, Javorník
  - Boehringer Ingelheim Investigational Site, Jeseník
  - Boehringer Ingelheim Investigational Site, Jicín
  - Boehringer Ingelheim Investigational Site, Jihlava
  - Boehringer Ingelheim Investigational Site, Jirkov
  - Boehringer Ingelheim Investigational Site, Kadaň
  - Boehringer Ingelheim Investigational Site, Kaplice
  - Boehringer Ingelheim Investigational Site, Karlovy Vary
  - Boehringer Ingelheim Investigational Site, Kladno
  - Boehringer Ingelheim Investigational Site, Klatovy
  - Boehringer Ingelheim Investigational Site, Klásterec N. Ohrí
  - Boehringer Ingelheim Investigational Site, Klobouky u Brna
  - Boehringer Ingelheim Investigational Site, Kolín
  - Boehringer Ingelheim Investigational Site, Konice
  - Boehringer Ingelheim Investigational Site, Kopřivnice
  - Boehringer Ingelheim Investigational Site, Kosmonosy
  - Boehringer Ingelheim Investigational Site, Kostelec nad Orlicí
  - Boehringer Ingelheim Investigational Site, Kralupy nad Vltavou
  - Boehringer Ingelheim Investigational Site, Králuv Dvur
  - Boehringer Ingelheim Investigational Site, Krnov
  - Boehringer Ingelheim Investigational Site, Kromeríz
  - Boehringer Ingelheim Investigational Site, Krouna
  - Boehringer Ingelheim Investigational Site, Krupka
  - Boehringer Ingelheim Investigational Site, Kunovice
  - Boehringer Ingelheim Investigational Site, Kuřim
  - Boehringer Ingelheim Investigational Site, Kyjov
  - Boehringer Ingelheim Investigational Site, Lanškroun
  - Boehringer Ingelheim Investigational Site, Ledec Nad Sázavou
  - Boehringer Ingelheim Investigational Site, Lenešice
  - Boehringer Ingelheim Investigational Site, Letohrad
  - Boehringer Ingelheim Investigational Site, Liberec
  - Boehringer Ingelheim Investigational Site, Liběšice
  - Boehringer Ingelheim Investigational Site, Libochovice
  - Boehringer Ingelheim Investigational Site, Lipová Lázne
  - Boehringer Ingelheim Investigational Site, Litoměřice
  - Boehringer Ingelheim Investigational Site, Litovel
  - Boehringer Ingelheim Investigational Site, Litvínov
  - Boehringer Ingelheim Investigational Site, Lomnice n.P.
  - Boehringer Ingelheim Investigational Site, Louny
  - Boehringer Ingelheim Investigational Site, Lovosice
  - Boehringer Ingelheim Investigational Site, Ludgérovice
  - Boehringer Ingelheim Investigational Site, Mariánské Lázne
  - Boehringer Ingelheim Investigational Site, Melník
  - Boehringer Ingelheim Investigational Site, Město Albrechtice
  - Boehringer Ingelheim Investigational Site, Milín
  - Boehringer Ingelheim Investigational Site, Milovice
  - Boehringer Ingelheim Investigational Site, Míretice
  - Boehringer Ingelheim Investigational Site, Mladá Boleslav
  - Boehringer Ingelheim Investigational Site, Mlázovice
  - Boehringer Ingelheim Investigational Site, Mnísek Pod Brdy
  - Boehringer Ingelheim Investigational Site, Modřice
  - Boehringer Ingelheim Investigational Site, Mohelnice
  - Boehringer Ingelheim Investigational Site, Mor.Budejovice
  - Boehringer Ingelheim Investigational Site, Mor.Krumlov
  - Boehringer Ingelheim Investigational Site, Mor.Nová Ves
  - Boehringer Ingelheim Investigational Site, Moravany
  - Boehringer Ingelheim Investigational Site, Most
  - Boehringer Ingelheim Investigational Site, Mýto
  - Boehringer Ingelheim Investigational Site, Nasavrky
  - Boehringer Ingelheim Investigational Site, Náchod
  - Boehringer Ingelheim Investigational Site, Námest Nad Oslavou
  - Boehringer Ingelheim Investigational Site, Nechanice
  - Boehringer Ingelheim Investigational Site, Neratovice
  - Boehringer Ingelheim Investigational Site, Nová Ves Pod Plesí
  - Boehringer Ingelheim Investigational Site, Nové Mesto Nad Metují
  - Boehringer Ingelheim Investigational Site, Nový Bor
  - Boehringer Ingelheim Investigational Site, Nový Bydzov
  - Boehringer Ingelheim Investigational Site, Nový Jicín
  - Boehringer Ingelheim Investigational Site, Nový Knín
  - Boehringer Ingelheim Investigational Site, Nymburk
  - Boehringer Ingelheim Investigational Site, Obrataň
  - Boehringer Ingelheim Investigational Site, Obríství
  - Boehringer Ingelheim Investigational Site, Olomouc
  - Boehringer Ingelheim Investigational Site, Opava
  - Boehringer Ingelheim Investigational Site, Opočno
  - Boehringer Ingelheim Investigational Site, Orlová
  - Boehringer Ingelheim Investigational Site, Ostrava
  - Boehringer Ingelheim Investigational Site, Otrokovice
  - Boehringer Ingelheim Investigational Site, Pacov
  - Boehringer Ingelheim Investigational Site, Pardubice
  - Boehringer Ingelheim Investigational Site, Pelhřimov
  - Boehringer Ingelheim Investigational Site, Petřvald
  - Boehringer Ingelheim Investigational Site, Pierov
  - Boehringer Ingelheim Investigational Site, Pilsen
  - Boehringer Ingelheim Investigational Site, Písek
  - Boehringer Ingelheim Investigational Site, Planá
  - Boehringer Ingelheim Investigational Site, Polná
  - Boehringer Ingelheim Investigational Site, Postoloprty
  - Boehringer Ingelheim Investigational Site, Postřelmov
  - Boehringer Ingelheim Investigational Site, Prachatice
  - Boehringer Ingelheim Investigational Site, Prague
  - Boehringer Ingelheim Investigational Site, Príbram
  - Boehringer Ingelheim Investigational Site, Prostějov
  - Boehringer Ingelheim Investigational Site, Přelouč
  - Boehringer Ingelheim Investigational Site, Přeštice
  - Boehringer Ingelheim Investigational Site, Radonice
  - Boehringer Ingelheim Investigational Site, Rakovník
  - Boehringer Ingelheim Investigational Site, Raspenava
  - Boehringer Ingelheim Investigational Site, Rícany U Brna
  - Boehringer Ingelheim Investigational Site, Rokycany
  - Boehringer Ingelheim Investigational Site, Roudnice nad Labem
  - Boehringer Ingelheim Investigational Site, Rožnov pod Radhoštěm
  - Boehringer Ingelheim Investigational Site, Ruda nad Moravou
  - Boehringer Ingelheim Investigational Site, Rudná U Prahy
  - Boehringer Ingelheim Investigational Site, Rumburk
  - Boehringer Ingelheim Investigational Site, Rychnov nad Kněžnou
  - Boehringer Ingelheim Investigational Site, Rýmarov
  - Boehringer Ingelheim Investigational Site, Řevnice
  - Boehringer Ingelheim Investigational Site, Semily
  - Boehringer Ingelheim Investigational Site, Senov U NJ
  - Boehringer Ingelheim Investigational Site, Skuteč
  - Boehringer Ingelheim Investigational Site, Slaný
  - Boehringer Ingelheim Investigational Site, Slatiňany
  - Boehringer Ingelheim Investigational Site, Slavicín
  - Boehringer Ingelheim Investigational Site, Slušovice
  - Boehringer Ingelheim Investigational Site, Smidary
  - Boehringer Ingelheim Investigational Site, Smiřice
  - Boehringer Ingelheim Investigational Site, Sokolov
  - Boehringer Ingelheim Investigational Site, Spálené Porící
  - Boehringer Ingelheim Investigational Site, Staré Mesto
  - Boehringer Ingelheim Investigational Site, Starý Plzenec
  - Boehringer Ingelheim Investigational Site, Stáhlavy
  - Boehringer Ingelheim Investigational Site, Stetí
  - Boehringer Ingelheim Investigational Site, Strakonice
  - Boehringer Ingelheim Investigational Site, Stríbro
  - Boehringer Ingelheim Investigational Site, Studená
  - Boehringer Ingelheim Investigational Site, Studénka
  - Boehringer Ingelheim Investigational Site, Svetlá Nad Sázavou
  - Boehringer Ingelheim Investigational Site, Šaratice
  - Boehringer Ingelheim Investigational Site, Štěnovice
  - Boehringer Ingelheim Investigational Site, Šumperk
  - Boehringer Ingelheim Investigational Site, Tábor
  - Boehringer Ingelheim Investigational Site, Teplice
  - Boehringer Ingelheim Investigational Site, Tišnov
  - Boehringer Ingelheim Investigational Site, Tlucná
  - Boehringer Ingelheim Investigational Site, Toužim
  - Boehringer Ingelheim Investigational Site, Trebíc
  - Boehringer Ingelheim Investigational Site, Tremosná
  - Boehringer Ingelheim Investigational Site, Trutnov
  - Boehringer Ingelheim Investigational Site, Třešť
  - Boehringer Ingelheim Investigational Site, Třinec
  - Boehringer Ingelheim Investigational Site, Tupesy
  - Boehringer Ingelheim Investigational Site, Turnov
  - Boehringer Ingelheim Investigational Site, Uherské Hradiste
  - Boehringer Ingelheim Investigational Site, Uherský Brod
  - Boehringer Ingelheim Investigational Site, Ústek
  - Boehringer Ingelheim Investigational Site, Ústí nad Labem
  - Boehringer Ingelheim Investigational Site, Ústí nad Orlicí
  - Boehringer Ingelheim Investigational Site, Val.Bystrice
  - Boehringer Ingelheim Investigational Site, Valasské Mezirící
  - Boehringer Ingelheim Investigational Site, Vamberk
  - Boehringer Ingelheim Investigational Site, Varnsdorf
  - Boehringer Ingelheim Investigational Site, Vápenná
  - Boehringer Ingelheim Investigational Site, Velká Bítes
  - Boehringer Ingelheim Investigational Site, Velké Mezirící
  - Boehringer Ingelheim Investigational Site, Velké Opatovice
  - Boehringer Ingelheim Investigational Site, Velké Porící
  - Boehringer Ingelheim Investigational Site, Veselí nad Moravou
  - Boehringer Ingelheim Investigational Site, Vintírov
  - Boehringer Ingelheim Investigational Site, Vlašim
  - Boehringer Ingelheim Investigational Site, Vodňany
  - Boehringer Ingelheim Investigational Site, Votice
  - Boehringer Ingelheim Investigational Site, Vrbno pod Pradědem
  - Boehringer Ingelheim Investigational Site, Vsetín
  - Boehringer Ingelheim Investigational Site, Vysoké Mýto
  - Boehringer Ingelheim Investigational Site, Vyškov
  - Boehringer Ingelheim Investigational Site, Zastávka
  - Boehringer Ingelheim Investigational Site, Zábieh
  - Boehringer Ingelheim Investigational Site, Zbýsov
  - Boehringer Ingelheim Investigational Site, Zdár Nad Sázavou
  - Boehringer Ingelheim Investigational Site, Zlín
  - Boehringer Ingelheim Investigational Site, Znojmo
  - Boehringer Ingelheim Investigational Site, Žamberk
  - Boehringer Ingelheim Investigational Site, Žatec
  - Boehringer Ingelheim Investigational Site, Žinkovy
  - Boehringer Ingelheim Investigational Site, Žirovnice
- Estonia (15):
  - Boehringer Ingelheim Investigational Site, Elva
  - Boehringer Ingelheim Investigational Site, Haapsalu
  - Boehringer Ingelheim Investigational Site, Jõhvi
  - Boehringer Ingelheim Investigational Site, Kohtla-Järve
  - Boehringer Ingelheim Investigational Site, Kose
  - Boehringer Ingelheim Investigational Site, Laane-Virumaa
  - Boehringer Ingelheim Investigational Site, Narva
  - Boehringer Ingelheim Investigational Site, Paide
  - Boehringer Ingelheim Investigational Site, Parne
  - Boehringer Ingelheim Investigational Site, Põlva
  - Boehringer Ingelheim Investigational Site, Rakvere
  - Boehringer Ingelheim Investigational Site, Sillamäe
  - Boehringer Ingelheim Investigational Site, Tallinn
  - Boehringer Ingelheim Investigational Site, Tartu
  - Boehringer Ingelheim Investigational Site, Viljandi
- Russia (13):
  - Boehringer Ingelheim Investigational Site, Bryansk
  - Boehringer Ingelheim Investigational Site, Dmitrov
  - Boehringer Ingelheim Investigational Site, Dolgoprudnii
  - Boehringer Ingelheim Investigational Site, Dzerzhinsk
  - Boehringer Ingelheim Investigational Site, Gukovscii
  - Boehringer Ingelheim Investigational Site, Ivanovo
  - Boehringer Ingelheim Investigational Site, Moscow
  - Boehringer Ingelheim Investigational Site, Nizhny Novgorod
  - Boehringer Ingelheim Investigational Site, Podolsk
  - Boehringer Ingelheim Investigational Site, Ryazan
  - Boehringer Ingelheim Investigational Site, Smolensk
  - Boehringer Ingelheim Investigational Site, Vladimir
  - Boehringer Ingelheim Investigational Site, Yaroslavl
- Slovakia (36):
  - Boehringer Ingelheim Investigational Site, Bardejov
  - Boehringer Ingelheim Investigational Site, Bánovce/Bebravou
  - Boehringer Ingelheim Investigational Site, Bošany
  - Boehringer Ingelheim Investigational Site, Bran?
  - Boehringer Ingelheim Investigational Site, Handlová
  - Boehringer Ingelheim Investigational Site, Humenné
  - Boehringer Ingelheim Investigational Site, Kežmarok
  - Boehringer Ingelheim Investigational Site, Kluknava
  - Boehringer Ingelheim Investigational Site, Košice
  - Boehringer Ingelheim Investigational Site, Krompachy
  - Boehringer Ingelheim Investigational Site, Liptovský Mikulás
  - Boehringer Ingelheim Investigational Site, Malacky
  - Boehringer Ingelheim Investigational Site, Martin
  - Boehringer Ingelheim Investigational Site, Michalovce
  - Boehringer Ingelheim Investigational Site, Námestovo
  - Boehringer Ingelheim Investigational Site, Nitra
  - Boehringer Ingelheim Investigational Site, Nove Mesto/Váhom
  - Boehringer Ingelheim Investigational Site, Pies?any
  - Boehringer Ingelheim Investigational Site, Poprad
  - Boehringer Ingelheim Investigational Site, Prešov
  - Boehringer Ingelheim Investigational Site, Ružomberok
  - Boehringer Ingelheim Investigational Site, Saint ?ubov?a
  - Boehringer Ingelheim Investigational Site, Se?ovská Polianka
  - Boehringer Ingelheim Investigational Site, Senec
  - Boehringer Ingelheim Investigational Site, Spisská Nová Ves
  - Boehringer Ingelheim Investigational Site, Stará Turá
  - Boehringer Ingelheim Investigational Site, Stropkov
  - Boehringer Ingelheim Investigational Site, Svinia
  - Boehringer Ingelheim Investigational Site, Topo??any
  - Boehringer Ingelheim Investigational Site, Torna?a
  - Boehringer Ingelheim Investigational Site, Trebišov
  - Boehringer Ingelheim Investigational Site, Tren?ín
  - Boehringer Ingelheim Investigational Site, Trhovište
  - Boehringer Ingelheim Investigational Site, Vranov/Top?ou
  - Boehringer Ingelheim Investigational Site, Vrútky
  - Boehringer Ingelheim Investigational Site, Žilina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number of patients:
  * treated set = 3569 (treated with Movalis)
  * full analysis set = 3473 (patients completed 2 visits and had baseline and final 12-item Short-Form Health Survey (SF12) score)
Groups:
- Meloxicam 7.5 mg Tablets, 15 mg Tablets or Injection: 7.5 - 15 mg once daily (intramuscular injection and/or tablet), depending on clinical need and judgement of physician
Period: Overall Study
Arm/Group | Meloxicam 7.5 mg Tablets, 15 mg Tablets or Injection
Started | 3569 (treated set = 3569 (treated with Movalis))
Completed | 3061 (Due to some missing termination information, the number of "completed" may be larger than 3061.)
Not Completed | 508
Not completed — Adverse Event | 18
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 1
Not completed — Missing termination information | 481
Not completed — Not specified reasons | 6

BASELINE CHARACTERISTICS:
Population: Treated set
Arm/Group | Meloxicam 7.5 mg Tablets, 15 mg Tablets or Injection
Number analyzed (Participants) | 3569
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13.8)
Sex/Gender, Customized [Number; unit: participants]
  Female | 2355
  Male | 1167
  Missing | 47

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Medical Outcomes Study 12-item Short-Form Health Survey, Version 2 Score From Baseline to Final Visit.
Description: Physical Component Summary (PCS) Mean Difference final-baseline score. The Medical Outcomes Study 12-item Short-Form Health Survey, version 2 (SF-12v2) was used as the instrument to measure any changes in physical wellbeing (physical component summary, PCS) and mental wellbeing (mental component summary, MCS) in patients taking MOVALIS® therapy for approximately 4 weeks. Worst value 0 (lowest wellbeing), best value 100 (highest wellbeing)
Time Frame: baseline and final visit (approximately 4 weeks)
Population: A total of 3569 patients from five Central and Eastern Europe (CEE) countries were entered in the study. These patients were treated with MOVALIS® therapy and formed the treated set (TS). Of these, 3473 patients completed two visits and had a baseline and final score for SF-12v2 and formed the full analysis set (FAS).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Meloxicam 7.5 mg Tablets, 15 mg Tablets or Injection
Number analyzed (Participants) | 3473
Units on a scale | 11.2 (9.5)

2. Primary Outcome: Mean Change in SF 12 MCS Score From Baseline to Final Final Visit.Medical Outcomes Study 12-Item Short-Form Health Survey, Version 2
Description: Mental Component Summary (MCS). Mean Difference final-baseline score. Worst value 0 (lowest wellbeing), best value 100 (highest wellbeing)
Time Frame: Baseline and final visit (approximately 4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Meloxicam 7.5 mg Tablets, 15 mg Tablets or Injection
Number analyzed (Participants) | 3473
Units on a scale | 6.2 (10.1)

3. Secondary Outcome: Change From Baseline of Pain Intensity on Visual Analogue Scale
Description: The effect of MOVALIS® on reduction of pain intensity was assessed by the change from baseline in patient assessment of pain intensity on a Visual Analogue Scale (VAS) ranging from 0 (no pain) to 100 (severe pain)
Time Frame: Approximately four weeks of treatment
Population: Full analysis set (FAS): This analysis was performed on all patients in FAS with available data on pain intensity on VAS at baseline and final visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Meloxicam 7.5 mg Tablets, 15 mg Tablets or Injection
Number analyzed (Participants) | 3459
Units on a scale | 41.9 (18.9)

4. Secondary Outcome: Patient Assessment of Efficacy
Description: Patient assessment of general efficacy of MOVALIS® using a 5-point scale (1 excellent; 2 very good; 3 good; 4 fair; 5 poor) was performed at visit 2.
  The patients have been placed into categories according to the points on a scale.
Time Frame: after approximately 4 weeks of treatment
Population: Full analysis set (FAS). This analysis was performed on all patients in FAS with available data on the global assessment of general efficacy.
Measure: Number; unit: Participants
Arm/Group | Meloxicam 7.5 mg Tablets, 15 mg Tablets or Injection
Number analyzed (Participants) | 3461
Participants
  Excellent | 803
  Very Good | 1540
  Good | 928
  Fair | 161
  Poor | 29

5. Secondary Outcome: Physician Assessment of Efficacy
Description: Physician assessment of general efficacy of MOVALIS® using a 5-point scale (1 excellent; 2 very good; 3 good; 4 fair; 5 poor) was performed at visit 2.
  The patients have been placed into categories according to the points on a scale.
Time Frame: after approximately 4 weeks of treatment
Population: Full analysis set (FAS): This analysis was performed on all patients in FAS with available data on physician assessment of efficacy.
Measure: Number; unit: Participants
Arm/Group | Meloxicam 7.5 mg Tablets, 15 mg Tablets or Injection
Number analyzed (Participants) | 3467
Participants
  Excellent | 879
  Very Good | 1652
  Good | 806
  Fair | 109
  Poor | 21

ADVERSE EVENTS:
Time Frame: 4 weeks + 5 days
Description: There were no serious adverse events (SAEs) nor AEs over 5% frequency reported
Arm/Group | Meloxicam 7.5 mg Tablets, 15 mg Tablets or Injection
Serious Adverse Events (participants affected / at risk) | 0/3569
Other Adverse Events (participants affected / at risk) | 0/3569

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.